CLINICAL TRIAL: NCT00308737
Title: Pulmonary Outcomes Within a 2-Year Period in Subjects With Diabetes Mellitus Treated With Technosphere /Insulin or Usual Antidiabetic Treatment and in Subjects Without Abnormalities in Glucose Control.
Brief Title: Safety of Inhaled Insulin With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-030
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes, Type 1; Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

ARMS (3):
- TI Inhalation Powder (Experimental): Technosphere® Insulin Inhalation Powder
  Interventions: Drug: Technosphere® Insulin Inhalation Powder
- Usual care (Other): Usual care
  Interventions: Drug: Usual Care
- Non-diabetes (No Intervention): Subjects without abnormalities in glucose control (Note: Hypoglycemia and HbA1c were not reported for this group)

INTERVENTIONS:
Drug: Technosphere® Insulin Inhalation Powder — Inhalation, 15U/30U
  Arms: TI Inhalation Powder
Drug: Usual Care — Subjects will receive antidiabetes treatment at the discretion of their physicians
  Arms: Usual care

SUMMARY:
Pulmonary Safety in Diabetics with T/I

ELIGIBILITY:
Inclusion Criteria:

* For All Subjects:

  * Nonsmoking
  * Body mass index <42 kg/m2
  * FEV1 greater than or equal to 70% of predicted , DLco and TLC greater than or equal to 80% of predicted at screening,
  * No abnormalities in screening pulmonary radiology
* For Subjects with diabetes mellitus:

  * Type 1 or type 2 diabetes for at least 2 years
  * HbA1c greater than or equal to 6.6 % and less than or equal to 12.0 %
* For Subjects without abnormalities in glucose control:

  * No history of diabetes
  * Normal results from a formal glucose tolerance test

Exclusion Criteria:

* History of chronic obstructive pulmonary disease, asthma, or other significant pulmonary disease
* Significant renal, hepatic, or cardiac disease
* Women who are pregnant, lactating, or planning on becoming pregnant
* Subjects who have participated in studies of other investigational drugs within the previous 3 months
* Evidence of severe complications of diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2053 (Actual)
Dates: Start 2005-06; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (175):
- United States (82):
  - Southwest Health Ltd Research Division, Phoenix, Arizona
  - Lovelace Scientific Resources, Phoenix, Arizona
  - Northwest Medical Center, Phoenix, Arizona
  - Arizona Center for Clinical Research, Phoenix, Arizona
  - Premiere Pharmaceutical Research LLC, Tempe, Arizona
  - Canyon Clinical Research, Tucson, Arizona
  - Arizona Research Associates, Tuscon, Arizona
  - Private Practice, Burlingame, California
  - Saint Agnes Medical Center, Fresno, California
  - Valley Research, Fresno, California
  - (Private Practice), Garden Grove, California
  - Diabetes/Lipid Management Center, Huntington Beach, California
  - Interlink Research Institute, Los Alamitos, California
  - Diabetes Care Center, Salinas, California
  - San Diego Sports Medicine and Family Health Center, San Diego, California
  - Dorothy L & James E Frank Diabetes Research Institute, San Mateo, California
  - Sansum Medical Research Institute, Santa Barbara, California
  - Encompass Clinical Research, Spring Valley, California
  - Kaiser Permanente, Denver, Colorado
  - Denver VA Medical Center, Denver, Colorado
  - Alliance Medical Group of Greater Waterbury, Middlebury, Connecticut
  - New Britain General Hosptal c?o Betsy Keller, New Britain, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Perimeter Institute for Clinical Research (PICR), Atlanta, Georgia
  - Executive Health and Research Associates Inc, Atlanta, Georgia
  - Rockdale Medical Research Associates, Conyers, Georgia
  - Private Practice, Decatur, Georgia
  - Atlanta Pharmaceutical Research Center, Dunwoody, Georgia
  - North Atlanta Endocrinology & Diabetes PC, Lawrenceville, Georgia
  - Southeastern Endocrine & Diabetes, Roswell, Georgia
  - Fox Valley Clinical Research Center LLC, Aurora, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Medical Research of Louisiana, Metairie, Louisiana
  - Ochsner Clinic and Foundation, New Orleans, Louisiana
  - Health Trends Research LLC, Baltimore, Maryland
  - Franklin Square Hospital, Baltimore, Maryland
  - MODEL Clinical Research, Towson, Maryland
  - East Coast Clinical Research Inc, Haverhill, Massachusetts
  - Clinical Research, Waltham, Massachusetts
  - Michigan Institute of Medicine, Livonia, Michigan
  - PPS Clinical Research / Southwest Medical Center, Chesterfield, Missouri
  - Healthcare Research, Florissant, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - MedEx Healthcare Research Inc, St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Billings Clinic Research Division, Billings, Montana
  - Your Doctors Care, Hillsborough, New Jersey
  - Hopewell Valley Family Medicine PA, Trenton, New Jersey
  - Umdnj-Som, Voorhees Township, New Jersey
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Lovelace Scientific Resources (Albuquerque), Albuquerque, New Mexico
  - Southwest Endocrinology Associates, Albuquerque, New Mexico
  - Physicians Associates of Park Place, Brooklyn, New York
  - Diabetes Care & Information Center of New York, Flushing, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - M.E.R.I., New York, New York
  - Physicians Clinical Research Service (PCRS) (SMO), White Plains, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Endocrine Research - Physician's East PA, Greenville, North Carolina
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Your Diabetes Endocrine Nutrition Group, Mentor, Ohio
  - New Hope Research of Oregon, Portland, Oregon
  - Buckingham Family Medicine, Doyleston, Pennsylvania
  - Bucks County Clinical Research, Morrisville, Pennsylvania
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Texas Familicare Clinical Research, Colleyville, Texas
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Medical Research Associates, Houston, Texas
  - North Texas Medical Research, Plano, Texas
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas
  - Scott & White Hospital and Clinic, Temple, Texas
  - McLennan County Medical Education and Research Foundation, Waco, Texas
  - Magna Center for Family Medicine, Magna, Utah
  - Davis Family Practice, Salt Lake City, Utah
  - Radiant Research Salt Lake City, Salt Lake City, Utah
  - Southeastern PA Med Inst LLC (SMO), Salt Lake City, Utah
  - Granger Medical Clinic, West Valley City, Utah
  - Hampton Roads Center for Clinical Research Inc, Norfolk, Virginia
  - Rainier Clinical Research Center Inc, Renton, Washington
  - Clinical Research Department Wenatchee Valley Medical Center, Wenatchee, Washington
- Canada (10):
  - Finchlea Medical Group, Brampton, Ontario
  - Courtice Health Centre, Courtice, Ontario, Ontario
  - Parkwood Hospital, London, Ontario
  - Quest Clinical Trials, Markham, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - The London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Lifestyle Metabolism Center, Thornhill, Ontario
  - Albany Medical Center, Toronto, Ontario
  - Lifestyle Metabolism Center (600-118 Eglinton Ave W), Toronto, Ontario
  - Manna Research, Toronto, Ontario
- Czechia (7):
  - Diabetologicka ambulance, Litoměřice, CZE
  - Surgery of Diabetology, Mělník, CZE
  - Diabetologicka a interni ambulance, Ostrava, CZE
  - Internal Clinic, Ostrava - Poruba, CZE
  - Diabetologicka a interni ambulance, Ostrava-Kunčice, CZE
  - Surgery of Diabetology Petrovice, Prague, CZE
  - FN Motol Interni Klinika, Prague, CZE
- Poland (14):
  - Klinika Endocrinologii Diabetologii I, Bialystock, POL
  - Oddzial Chorob Wewnetrznych, Bialystock, POL
  - Dzial Badan Klinicznych Malopoiskie, Krakow, POL
  - Endokrynologiczno Metaboliczne DIAB_ENDO_MET, Krakow, POL
  - III Oddzial Chorob Wewnetrznych Szpital, Krakow, POL
  - Oddzial Wewnetrzny B, Lodz, POL
  - Klliniczny nr 1 im Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz, POL
  - Oddzial Diabetologiczny Centrum, Lodz, POL
  - Spzital Kolejowy imm Wlodzimierza Roeflera, Pruszków, POL
  - Klinika Medycyny Rodzinnej i Chorob, Warsaw, POL
  - Katedra i Klinika Gastroentereologii i, Warsaw, POL
  - Oddzial Chorob Wewnetznych i Diabetologii, Warsaw, POL
  - ZPZOZ w Otwocku Szpital Miejski, Warsaw, POL
  - Oddzial Internistyczny Specjalistyczna, Łask, POL
- Russia (25):
  - Kemerovo State Medical Academy of Ministry of Health, Kemerovo, RUS
  - NHI Kemerovo Regional Clinical Hospital, Kemerovo, RUS
  - NI Principal Military Clinical Hospital n a academician N.N. Burdenko of the Ministry of Defense, Moscow, RUS
  - Russian State Medical University City Hospital # 4, Moscow, RUS
  - NI Endrocrinological Research Centre of RAMS In patient replacing technologies department, Moscow, RUS
  - Russian Academy of Medical Sciences National Research Ctr for Endocrinology Institute of Diabetes, Moscow, RUS
  - Russian State Medical University Central Clinical Hospital Russian Science Academy, Moscow, RUS
  - RAAMS Endocrinology and Diabetology Department, Moscow, RUS
  - SIH of Moscow City Clinical Hopsital #81 Endocrinology and Diabetology, Moscow, RUS
  - NI Moscow Regional Scientific Research Clinical Institute na MF Vladimirsky, Moscow, RUS
  - Municipal Clinical Hospital #13, Moscow, RUS
  - Moscow State Medical-Stomatological University City Clinical Hospital # 23, Moscow, RUS
  - Ryazan State Medical University na academician IP Pavlov, Ryazan, RUS
  - Krestovsky Island Medical Institute, Saint Petersburg, RUS
  - St Petersburg NHI City Polytclinic #77 City Diabetological Center #4, Saint Petersburg, RUS
  - Central Medical Sanitary Unit #122, Saint Petersburg, RUS
  - St Petersburg NHI Municipal Multi-Speciality Hospital # 2, Saint Petersburg, RUS
  - St Petersburg Medical Academy St Elizabeth Hospital, Saint Petersburg, RUS
  - Pavlov State Medical Univ of St Petersburg, Saint Petersburg, RUS
  - NEI HPE Smolensk State Medical Academy of FAHSD RNHI Smolensk Regional Clinical Hospital, Smolensk, RUS
  - Clinical Pharm Dept of Yaroslavl Clin Hospital, Yaroslavl, RUS
  - MHI Clinical Hospital for Emergency Care na NV Soloviev, Yaroslavl, RUS
  - NHI Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS
  - Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS
  - Federal State Institution Pulmonology Research Institute of Federal Agency of HC&SD, Moscow
- Spain (7):
  - Fundacio Sarda Farriol, Barcelona, ESP
  - Fundacion Jimenez Diaz Servicio Endocrinologia y Nutricion, Madrid, ESP
  - Hospital 12 de Octubre Consultas Extremas - Endocrinologia, Madrid, ESP
  - Hospital Universitario de la Paz, Madrid, ESP
  - Seville, ESP
  - Hospital Univ Virgen del Rocío Scio Endocrinología Centro de Diagnosticos Pl Baja, Seville, ESP
  - Hospital Clinic I Provincial, Barcelona
- Ukraine (18):
  - Bukovinian State Medical University Dept of Clinical Immun, Chernivtcy, UKR
  - Dniepropetrovsh State Medical Academy, Dniepropetrovsk, UKR
  - Donetsk State Medical University, Donetsk, UKR
  - Railway Clinical Hospital on Donetsk Station, Donetsk, UKR
  - V Danilevsky Inst of Endocrinology Pathology, Kharkiv, UKR
  - Medical University at Kiev Center of Endocrinology and Metab, Kiev, UKR
  - Chair Family Med of National Med University, Kiev, UKR
  - Ukr Scientifically Practical Centre of Endocrine Surgery, Kiev, UKR
  - Lugansk State Medical University Chair of Hosp Therapy #2, Luhansk, UKR
  - Lugansk State Medical University Chair of Therapy #1, Luhansk, UKR
  - Chair of Endocrin & Clinical Pharmacology of Lvov State Medical University, Lviv, UKR
  - Odessa State Medical University Dept of Gen Practice and Med Rehab, Odesa, UKR
  - Odessa Reg. Clinical Hosp Outpatient Department, Odesa, UKR
  - Odessa State Med Dept of Family Med and Gen Practice, Odesa, UKR
  - Crimean State Medical University Dept of Therapy #1, Simferopol, UKR
  - Vinnitsa State Medical University, Vinnitsa, UKR
  - Outpatient Clinic of Family Physician "Rusanovka", Kiev
  - Public Institution City Policlinic #20 Odessa, Odesa
- United Kingdom (12):
  - Barnsley Hospital, Barnsley, GBR
  - Kingthorne Group Practice, Doncaster, GBR
  - Manny Cussins Centre, Leeds, GBR
  - Royal liverpool University Hospital, Liverpool, GBR
  - Clinical Research Centre The Royal London Hospital, London, GBR
  - Medinova Research Mount Vernon Hospital, Middlesex, GBR
  - Edith Cavel Hospital Diabetes Centre, Peterborough, GBR
  - Northern General Hospital, Sheffield, GBR
  - Woolpit Medical Practice, Suffolk, GBR
  - West Suffolk Hospital, Suffolk, GBR
  - Birmingham Heartland Hospital, West Midlands, GBR
  - Bradford Hospital Dept of Diabetes & Endocrinology, West Yorkshire, GBR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled July 25, 2005 Multi-national trial conducted in Canada, Czech Republic, Poland, Russia, Spain, Ukraine, UK, and US
Pre-assignment Details: Subjects were required to meet all inclusion/exclusion criteria 3741 screened/2053 eligible of which all were randomized, including 164 non-diabetics - 1688 screen failures
  17 diabetics randomized but not dosed
  1 non-diabetic elected not to participate
Groups:
- Technosphere® Insulin: Technosphere Insulin with or without basal insulin, or oral anti-diabetic medications, or any combination of the previous.
- Usual Care: Usual care may consist of oral anti-diabetic medications, basal insulin, subcutaneous prandial insulin, or any combination of the previous.
- Non-diabetes: Subjects without abnormalities in glucose control
Period: Overall Study
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Started | 938 | 951 | 164
Completed | 475 | 662 | 127
Not Completed | 463 | 289 | 37
Not completed — Adverse Event | 104 | 9 | 0
Not completed — Death | 4 | 3 | 0
Not completed — Lost to Follow-up | 56 | 80 | 5
Not completed — Physician Decision | 15 | 2 | 1
Not completed — Protocol Violation | 34 | 9 | 5
Not completed — Withdrawal by Subject | 218 | 166 | 18
Not completed — Various | 32 | 20 | 8

BASELINE CHARACTERISTICS:
Population: Safety population, excluding subjects who were not dosed with study medication (17 diabetics randomized but not dosed, 1 non-diabetic elected not to participate)
Groups:
- Technosphere® Insulin: Technosphere Insulin
- Total: Total of all reporting groups
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes | Total
Number analyzed (Participants) | 923 | 949 | 163 | 2035
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.55) | 50.4 (11.62) | 38.2 (12.59) | 49.6 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 366 | 371 | 92 | 829
  Male | 557 | 578 | 71 | 1206
Body mass index [Mean (Standard Deviation); unit: kilograms per meter squared] — Body mass index
  kilograms per meter squared | 29.87 (5.366) | 29.76 (5.035) | 25.27 (4.494) | 29.5 (5.29)
HbA1c [Mean (Standard Deviation); unit: percentage] — Glycated hemoglobin
  percentage | 8.7 (1.39) | 8.7 (1.38) | 0 (0) | 8.4 (1.61)
Weight [Mean (Standard Deviation); unit: kilograms] — Weight in kilograms
  kilograms | 87.69 (18.628) | 87.53 (17.638) | 74.35 (16.204) | 86.6 (18.33)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 24 in Forced Expiratory Volume in 1 Second (FEV1) by MMRM for TI vs Usual Care
Description: Change from Baseline to End of Study in FEV1 by MMRM
Time Frame: Baseline to Month 24
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Technosphere® Insulin | Usual Care
Number analyzed (Participants) | 730 | 824
liters | -0.16 (0.208) | -0.12 (0.211)
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Mixed model repeated measures with fixed effects diabetes type, visit, pooled site and treatment and baseline FEV1 as a covariate; Test type: Non-Inferiority or Equivalence — Comparison of TI + Usual Care to Usual Care only; Mixed Models Analysis; Repeated measures; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [0.014 to 0.060]

2. Secondary Outcome: Change From Baseline to Last Measurement in FEV1 for TI vs Usual Care
Description: Change from Baseline to last measurement(Month 24) in FEV1
Time Frame: Baseline to Month 24
Population: Intention to Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | Technosphere® Insulin | Usual Care
Number analyzed (Participants) | 730 | 824
liters | -0.128 [-0.144 to -0.113] | -0.092 [-0.107 to -0.077]
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; ANCOVA model with treatment site, diabetes type, and baseline FEV1; Test type: Non-Inferiority or Equivalence — The null hypothesis tested was that the FEV1 change from Baseline for the TI group is no greater than 50 mL/year above the change in the usual care treatment group. Assuming SD of 100 mL/y, 80% power, and 5% (1-tailed) significance level, it was determined that 50 subjects were required for each of the diabetes treatment groups. Final sample size was selected for the incidence of a >= 15% decrease in FEV1 end point; ANCOVA; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [0.016 to 0.057]

3. Secondary Outcome: Change From Baseline to Month 24 in Forced Vital Capacity (FVC) by MMRM
Description: Change from Baseline to Month 24 in FVC by MMRM
Time Frame: Baseline to Month 24
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Number analyzed (Participants) | 730 | 824 | 145
liters | -0.14 (0.242) | -0.11 (0.262) | -0.09 (0.210)
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Mixed model repeated measures with fixed effects diabetes type, visit, pooled site and treatment and baseline FVC as a covariate; Test type: Superiority or Other; Mixed Models Analysis; Repeated measures; Mean Difference (Net) = 0.034, 95% CI 2-sided [0.008 to 0.061]

4. Secondary Outcome: Change From Baseline to Month 24 in Total Lung Capacity (TLC) by MMRM
Description: Change from baseline to Month 24 in TLC by MMRM
Time Frame: Baseline to Month 24
Population: participants in ITT population with available data
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Number analyzed (Participants) | 717 | 817 | 144
liters | -0.05 (0.321) | -0.07 (0.322) | -0.02 (0.297)
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Mixed model repeated measures with fixed effects diabetes type, visit, pooled site, and treatment and baseline TLC as a covariate; Test type: Superiority or Other; Mixed Models Analysis; Repeated measures; Mean Difference (Net) = -0.005, 95% CI 2-sided [-0.042 to 0.031]

5. Secondary Outcome: Change From Baseline to Month 24 in Hemoglobin Corrected DLco by MMRM
Description: Change from baseline to Month 24 in hemoglobin-corrected DLco by MMRM
Time Frame: Baseline to Month 24
Population: participants in ITT population with available data
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Number analyzed (Participants) | 723 | 818 | 144
mL/min/mmHg | -1.60 (2.830) | -1.36 (2.862) | -1.33 (3.203)
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Repeated measures; Mean Difference (Net) = 0.269, 95% CI 2-sided [-0.037 to 0.574]

6. Secondary Outcome: Forced Vital Capacity (FVC) Decrease of ≥ 15% From Baseline Value at Last Measurement
Description: FVC Decrease of ≥15% from Baseline Value at Last Measurement
Time Frame: Baseline to Month 24
Population: participants in ITT population with available data
Measure: Number; unit: participants
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Number analyzed (Participants) | 730 | 824 | 145
participants | 23 | 17 | 2
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Logistic regression excluding non-diabetics; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.6475, 95% CI 2-sided [0.3432 to 1.2219]

7. Secondary Outcome: Total Lung Capacity (TLC) Decrease of ≥ 15% From Baseline Value at Last Measurement
Description: TLC Decrease of ≥ 15% from Baseline Value at Last Measurement
Time Frame: Baseline to Month 24
Population: participants in ITT population with available data
Measure: Number; unit: Participants
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Number analyzed (Participants) | 717 | 817 | 144
Participants | 7 | 6 | 1
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Logistic regression excluding non-diabetics; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.7504, 95% CI 2-sided [0.2510 to 2.2431]

8. Secondary Outcome: Hemoglobin-Corrected Diffusing Capacity of the Lung for Carbon Monoxide (DLco) Decrease of ≥ 15% From Baseline Value at Last Measurement
Description: Hemoglobin-corrected DLco decrease of ≥ 15% from baseline value at last measurement
Time Frame: Baseline to Month 24
Population: participants in ITT population with available data
Measure: Number; unit: Participants
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Number analyzed (Participants) | 723 | 818 | 144
Participants | 105 | 108 | 20
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Logistic regression excluding non-diabetics; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.8953, 95% CI 2-sided [0.6703 to 1.1958]

9. Secondary Outcome: Hemoglobin-Corrected Diffusing Capacity of the Lung for Carbon Monoxide (DLco) Decrease of >3 ml/Min/mmHg From Baseline Value at Last Measurement
Description: Hemoglobin-corrected DLco decrease of >3 ml/min/mmHg from baseline value at last measurement
Time Frame: Baseline to Month 24
Population: participants in ITT population with available data
Measure: Number; unit: Participants
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Number analyzed (Participants) | 723 | 818 | 144
Participants | 181 | 181 | 40
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Logistic regression excluding non-diabetics; Test type: Superiority or Other; Regression, Logistic; Odds Ratio, log = 0.8509, 95% CI 2-sided [0.6722 to 1.0770]

10. Secondary Outcome: Change From Baseline in Glycated Hemoglobin A1c (HbA1c) at Last Measurement for TI vs Usual Care
Description: Change from baseline in HbA1c at last measurement
Time Frame: Baseline to Month 24
Population: Intention to treat (ITT) with last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Technosphere® Insulin | Usual Care
Number analyzed (Participants) | 725 | 818
percentage | -0.42 (1.410) | -0.49 (1.37)

11. Secondary Outcome: Change in Weight From Baseline at Month 24
Description: Change from baseline in weight at Month 24
Time Frame: Baseline to Month 24
Population: Safety population at Month 24
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Number analyzed (Participants) | 185 | 664 | 126
kilograms | 1.0 (6.653) | 1.64 (5.066) | 1.19 (4.457)
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Two sample t-test; Test type: Superiority or Other; p = 0.112, t-test, 2 sided

12. Primary Outcome: FEV1 Decrease of ≥ 15% From Baseline Value at Last Measurement for TI vs Usual Care
Description: FEV1 decrease of ≥ 15% from Baseline value at last measurement
Time Frame: Baseline to Month 24
Population: Intention to Treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Technosphere® Insulin | Usual Care
Number analyzed (Participants) | 730 | 824
Participants | 42 | 27
Statistical Analysis 1: Comparison: Technosphere® Insulin vs Usual Care; Logistic regression excluding non-diabetics; Test type: Non-Inferiority or Equivalence — The null hypothesis tested was that the difference in incidence of a decrease of ≥ 15% in FEV1 between the treatment groups not be greater than 5% for TI when compared with the usual care treatment group. Assuming an incidence rate of 15% for FEV1 and a noninferiority criterion of a 5% difference in incidence between the treatment groups, approximately 625 subjects per group were required for 80% power and an alpha of 5% (1 tailed); Regression, Logistic; Odds Ratio (OR) = -2.4767, 95% CI 2-sided [-4.5578 to -0.3956]

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- Usual Care: Usual care (taking insulin)
Arm/Group | Technosphere® Insulin | Usual Care | Non-diabetes
Serious Adverse Events (participants affected / at risk) | 92/923 | 91/949 | 5/163
Other Adverse Events (participants affected / at risk) | 559/923 | 472/949 | 47/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Technosphere® Insulin (N=923) | Usual Care (N=949) | Non-diabetes (N=163)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 5 | 3 | 0
Myocardial infarction (Cardiac disorders) | 2 | 4 | 0
Angina unstable (Cardiac disorders) | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Coronary artery atherosclerosis (Cardiac disorders) | 1 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 2 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 3 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Benign colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 2 | 0 | 0
Generalised oedema (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 4 | 0
Diabetic gangrene (Infections and infestations) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0 | 0
Cellulitis streptococcal (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0
Injection site cellulitis (Infections and infestations) | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Postoperative infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Staphylococcal scalded skin syndrome (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 10 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 6 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 | 0 | 0
Ketosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 5 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 4 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 2 | 0
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 3 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Atherosclerosis obliterans (Vascular disorders) | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Technosphere® Insulin (N=923) | Usual Care (N=949) | Non-diabetes (N=163)
Upper respiratory tract infection (Infections and infestations) | 119 | 143 | 35
Nasopharyngitis (Infections and infestations) | 67 | 69 | 14
Hypoglycaemia (Metabolism and nutrition disorders) | 365 | 370 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 257 | 42 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.